CLINICAL TRIAL: NCT02410317
Title: Ropivacaine Through Continuous Infusion Versus Epidural Morphine for Postoperative Analgesia After Emergency Cesarean Section
Acronym: ROMANCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Eudract 2014-002044-41
Record Dates: First submitted 2015-04-01; First posted 2015-04-07 (Estimated); Last update posted 2022-11-08 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain; Postoperative morphine consumption; Emergency cesarean delivery; Ropivacaine; Local anesthetic wound 48-hours infusion; Emergency cesarean section
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Morphine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous wound infusion group (Experimental): Patients receive analgesia through a multiorifice wound catheter connected to ropivacaine infusion. Saline solution is given in the epidural bolus.
  Interventions: Drug: Ropivacaine
- Epidural morphine group (Active Comparator): Patients receive epidural analgesia through an epidural bolus of morphine. Saline solution is perfused through the wound catheter.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Ropivacaine
  Arms: Continuous wound infusion group
Drug: Morphine
  Arms: Epidural morphine group

SUMMARY:
The cesarean section is one of the most commonly performed surgeries in the world and it represents 20% of the births in France. Postoperative pain is moderate-to-severe during the first 48 hours after this procedure. Thereby its control is prominent for the medical team in order to shorten the duration of hospital stay as well as to permit an early return to daily activities for these surgical patients.

Pain control after cesarean section is usually based on non-opioids and epidural administration of morphine if an epidural catheter has been previously placed for the procedure. However epidural morphine is associated with a number of side effects. Wound infiltration with local anesthetics has been widely used in the multimodal management of postoperative pain and it may reduce postoperative morphine consumption.

In patients enrolled for emergency cesarean delivery with epidural catheter, the objective of this study will be to compare the analgesia provided by a local anesthetic wound 48-hours infusion through a multiorifice catheter (ropivacaine 2 mg/mL) versus epidural analgesia (epidural morphine bolus). Quality of pain control will be assessed with the measurements of morphine consumption and pain scores at rest and during mobilisation over 48 hours. At 3 months, patients will be interviewed to assess their residual pain and their satisfaction.

It is hypothesized that local anesthetic wound infusion would be non-inferior than epidural morphine analgesia to control pain after cesarean section, and be associated with a reduction of side effects related to the analgesics.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age 18 years
* ASA-1 and 2 Parturient
* Emergency Cesarean delivery under epidural anesthesia
* Suprapubic incision used for cesarean section
* Functional epidural Catheter before the cesarean decision

(ASA Scores : Physical Status score)

Exclusion Criteria:

* ASA-3 and 4 Parturient
* BMI > 35 (before pregnancy)
* Existing chronic pain
* Contra-indication to study treatments
* Chronic use of analgesics or morphinic
* Preeclampsia
* Infection
* < 37 weeks pregnant +/- 3 days

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2021-08-28 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Pain score during mobilization | at 24 hours
  Visual analog scale for pain while the patient moves from lying to sitting

SECONDARY OUTCOMES:
Pain score at rest | at 2, 6(+/-1h), 12(+/-1h), 24(+/-2h), and 48 hours (+/-3h)
  Visual analog scale for pain while the patient is at rest
Pain score during mobilization | at 2, 6(+/-1h), 12(+/-1h), 24(+/-2h), and 48 hours (+/-3h)
  Visual analog scale for pain while the patient moves from lying to sitting
The incidence of morphine side effects: nausea, vomiting, pruritus | at 2, 6(+/-1h), 12(+/-1h), 24(+/-2h), and 48 hours (+/-3h)
  At every time points, side effects will be recorded
Duration of Indwelling Urethral Catheters | at 2, 6(+/-1h), 12(+/-1h), 24(+/-2h), and 48 hours (+/-3h)
  At ever time points, the presence of urethral catheter will be recorded and total duration will be compared.
Recovery of bowel function | at 2, 6(+/-1h), 12(+/-1h), 24(+/-2h), and 48 hours (+/-3h)
  At ever time points, patients will be asked whether they recovered bowel function and total duration to recover bowel function will be compared.
Morphine consumption dose | During hospital stay (an average of 3 days)
  Total dose of morphine consumed for pain management after the epidural bolus
Parturient satisfaction score | at 48 hours
  Satisfaction about pain management and breastfeeding
Complications during wound-catheter removal | at 48 hours
  Fever, pain, difficulties and infection at removal
Delay between birth and breastfeeding | During hospital stay (an average of 3 days)
Duration of stay | Hospital stay (an average of 3 days)
Residual pain | 3 months
  Numeric Rating Scale for Pain by phone interview

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Couple Enfant - CHU de Grenoble, Grenoble, France

REFERENCES:
- [Background] Fuller JG, McMorland GH, Douglas MJ, Palmer L. Epidural morphine for analgesia after caesarean section: a report of 4880 patients. Can J Anaesth. 1990 Sep;37(6):636-40. doi: 10.1007/BF03006481. PMID 2208533
- [Background] Palmer CM, Nogami WM, Van Maren G, Alves DM. Postcesarean epidural morphine: a dose-response study. Anesth Analg. 2000 Apr;90(4):887-91. doi: 10.1097/00000539-200004000-00021. PMID 10735794
- [Background] Bamigboye AA, Hofmeyr GJ. Local anaesthetic wound infiltration and abdominal nerves block during caesarean section for postoperative pain relief. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD006954. doi: 10.1002/14651858.CD006954.pub2. PMID 19588413
- [Background] Mecklem DW, Humphrey MD, Hicks RW. Efficacy of bupivacaine delivered by wound catheter for post-Caesarean section analgesia. Aust N Z J Obstet Gynaecol. 1995 Nov;35(4):416-21. doi: 10.1111/j.1479-828x.1995.tb02156.x. PMID 8717568
- [Background] Ranta PO, Ala-Kokko TI, Kukkonen JE, Ohtonen PP, Raudaskoski TH, Reponen PK, Rawal N. Incisional and epidural analgesia after caesarean delivery: a prospective, placebo-controlled, randomised clinical study. Int J Obstet Anesth. 2006 Jul;15(3):189-94. doi: 10.1016/j.ijoa.2006.02.003. PMID 16798442
- [Background] O'Neill P, Duarte F, Ribeiro I, Centeno MJ, Moreira J. Ropivacaine continuous wound infusion versus epidural morphine for postoperative analgesia after cesarean delivery: a randomized controlled trial. Anesth Analg. 2012 Jan;114(1):179-85. doi: 10.1213/ANE.0b013e3182368e87. Epub 2011 Oct 24. PMID 22025490
- [Background] Siddik SM, Aouad MT, Jalbout MI, Rizk LB, Kamar GH, Baraka AS. Diclofenac and/or propacetamol for postoperative pain management after cesarean delivery in patients receiving patient controlled analgesia morphine. Reg Anesth Pain Med. 2001 Jul-Aug;26(4):310-5. doi: 10.1053/rapm.2001.21828. PMID 11464348
- [Background] Rackelboom T, Strat SL, Silvera S, Schmitz T, Bassot A, Goffinet F, Ozier Y, Beaussier M, Mignon A. Improving continuous wound infusion effectiveness for postoperative analgesia after cesarean delivery: a randomized controlled trial. Obstet Gynecol. 2010 Oct;116(4):893-900. doi: 10.1097/AOG.0b013e3181f38ac6. PMID 20859153